CLINICAL TRIAL: NCT03217669
Title: Phase I Study of Epacadostat (INCB24360) in Combination With Sirolimus in Advanced Malignancy
Brief Title: Epacadostat (INCB24360) in Combination With Sirolimus in Advanced Malignancy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chao Huang (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Sponsor-Investigator, Chao Huang, Medical Doctor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2016-Epacadostat+SIRO
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Tumor; Non-small Cell Lung Cancer (NSCLC)
Keywords: epacadostat; sirolimus
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — epacadostat; Sirolimus

STUDY DESIGN:
Intervention Model Description: For the Dose Escalation cohort: Traditional 3+3 dose escalation design. For the Dose Expansion cohort: Once recommended phase two dose (RP2D) is defined by the PI, a total of 10 NSCLC patients who meet eligibility will be enrolled in the dose expansion cohort. If RP2D is not defined for any reason, the study will be terminated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sirolimus/Epacadostat Dose Escalation (Experimental): Traditional 3 + 3 dose escalation design.
  Starting doses: sirolimus 3milligrams (mg) loading/1mg maintenance and epacadostat 300mg twice daily (BID). If 0 in 3 subjects develops dose limiting toxicity (DLT), next 3 subjects will be treated at dose level 2 (DL2): sirolimus 6mg loading/2mg maintenance and epacadostat 300mg BID. If 1 subject in dose level 1 (DL1) develops DLT, 3 additional subjects will be enrolled in DL1. If 2 or more subjects in a total of 6 subjects, or 2 or more subjects in the initial 3 subjects develop DLT, the next 3 subjects will be treated at dose level -1 (DL-1): 3mg loading/1mg sirolimus + epacadostat 100mg BID. If only 1 subject in a total of 6 develops DLT, dose escalation to DL2 will be made for the next 3 subjects. Same algorithm will apply to DL2 except no further dose escalation/de-escalation will be made.
  Sirolimus lead-in phase: loading dose on day -7 and maintenance dose starting day -6. On Cycle 1 Day 1, epacadostat 300mg BID will be added.
  Interventions: Drug: Epacadostat; Drug: sirolimus
- Sirolimus/Epacadostat Dose Expansion (Experimental): Once recommended phase 2 dose (RP2D) is defined, a total of 10 non-small cell lung cancer (NSCLC) patients who meet eligibility will be enrolled in the dose expansion cohort. Treatment will be sirolimus RP2D once daily and epacadostat RP2D twice daily (BID).
  Sirolimus lead-in phase: loading dose on day -7 and maintenance dose starting day -6. On Cycle 1 Day 1, epacadostat 300mg BID will be added.
  Interventions: Drug: Epacadostat; Drug: sirolimus

INTERVENTIONS:
Drug: Epacadostat — Epacadostat tablet: 100mg or 300mg
  Other Names: INCB24360
Drug: sirolimus — Sirolimus tablet: 1mg, 2mg, 3mg, or 6mg
  Other Names: rapamycin; rapamune

SUMMARY:
This is a small phase I study with dose escalation and dose expansion cohorts. The former cohort will need up to 12 subjects with advanced solid tumor to define feasibility and recommended phase 2 dose (RP2D); the latter up to 10 subjects to further define safety. Study subjects will be adults with advanced solid tumor (dose escalation) and advanced non-small cell lung cancer (NSCLC) who progressed on at least one first-line systemic therapy (dose expansion).

DETAILED DESCRIPTION:
Indoleamine 2,3 dioxygenase-1 (IDO1) is a target of cancer immunotherapy. Epacadostat (INCB24360) is an oral IDO1 inhibitor. IDO1 activation blocks T-cell activation, enhances T-cell apoptosis and promotes the differentiation of naïve T cells to regulatory T cells (Tregs). Preclinical findings suggest that IDO1 is critical for cancers to evade immune surveillance and can be exploited for cancer immunotherapy.

Sirolimus is an oral Mammalian Target Of Rapamycin (mTOR) inhibitor. Protein Kinase B mTOR pathway has been considered one of major signaling cascade downstream of receptor kinases in human cells. Its activation in human cancer cells prompted scientists to develop its inhibitors.

Preclinical findings found that sirolimus can enhance activity of anti-Programmed Death-1 (PD-1) antibody by suppressing Programmed Death Ligand-1 (PD-L1) expression in human lung cancer models. Sirolimus is also known to suppress function of Tregs which contribute to immune evasion in cancer.

Other research groups also reported that autophagy is essential for Thymus cell/lymphocyte (T-cell) -mediated apoptosis which can be enhanced by AKT/mTOR/Phosphoinositide 3-kinase (PI3K) inhibitors. These studies indicate that autophagy is essential for T-cell mediated apoptosis signaling. Because autophagy is at least partially down-regulated by mTOR, mTOR inhibitors such as sirolimus can be used to pharmacologically induce autophagy. Overall, these findings suggest that activation of mTOR and resultant suppression of autophagy play a critical role in resistance of IDO1 inhibitor.

There is a clear unmet need for patients with advanced NSCLC whose median survival is approximately one year. Those who progressed on both standard first-line chemotherapy and second line anti-PD-1 inhibitor do not have any standard therapeutic option. Novel therapeutic strategy needs to develop for this population.

The IDO1 inhibitor epacadostat is currently being investigated in clinical trials in combination with various agents. However, these existing studies do not consider that mTOR and/or autophagy are key mechanisms of its resistance despite the abovementioned background information. The purpose of this phase I study is to test the combination of sirolimus with the IDO1 inhibitor in order to overcome potential resistance mechanisms associated with the use of IDO1.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the inclusion criteria to participate in this study.

* Ability to understand and the willingness to sign a written informed consent.
* Prior treatment with at least one line of systemic therapy.
* Dose escalation: subjects with advanced and unresectable solid tumor who progressed on at least one line of systemic therapy, and no approved therapy or standard therapy with demonstrated clinical benefit exists; and all subjects with T790M mutation positive NSCLC have progressed on osimertinib.

  *Note - Disease measurability is not required for dose escalation.
* Dose expansion: subjects with metastatic or recurrent NSCLC who progressed on at least one line of systemic therapy for metastatic or recurrent disease, which must include anti PD-1 or PD-L1 inhibitor, and must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and accessible tumor for biopsy. Molecular status of Epidermal Growth Factor Receptor (EGFR) and Anaplastic Lymphoma Kinase (ALK) must have been assessed for nonsquamous NSCLC. Those with activating EGFR mutation or ALK gene arrangement must have progressed on at least one kinase inhibitor.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status #0-2.
* Adequate organ and marrow function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/microliter (mcL)
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9 grams per deciliter (g/dL)
  * Total bilirubin within normal institutional limits
  * Aspartate Aminotransferase (AST) Serum Glutamic Oxaloacetic Transaminase (SGOT) ≤ 2.5 X institutional upper limit of normal (ULN)
  * Alanine Aminotransferase (ALT) Serum Glutamic Pyruvic Transaminase (SPGT) ≤ 2.5 X ULN
  * Alkaline Phosphatase Level (ALP) ≤ 2.5 X ULN
  * Serum creatinine ≤ 1.5 X ULN or Creatinine Clearance (CrCl) ≥ 50ml/min
  * Note: Subjects with bone metastasis and no liver metastasis on screening image may enroll if ALP is <5 X ULN. Subjects with liver metastasis may enroll if all of AST/ALT/ALP are <5 X ULN. However, subjects with extensive liver metastasis occupying more than 50% of liver parenchyma will be excluded.
  * Activated partial thromboplastin time (aPTT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy, as long as partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants.
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

  * A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)

Exclusion Criteria:

Participants meeting any of the exclusion criteria at baseline will be excluded from study participation.

* Current or anticipated use of other investigational agents while participating in this study.
* Participation in any other study in which receipt of an investigational study drug occurred within 28 days or 5 half-lives (whichever is longer) before first dose.
* Subjects who have received an IDO inhibitor. Subjects who have received other immune checkpoint inhibitors (e.g. anti-PD-1, anti-PD-L1, and any other treatment targeting T-cell) will be permitted. Subjects who have received experimental vaccines or other immune therapies should be discussed with the Principal Investigator (PI) to confirm eligibility.
* Subjects who have received sirolimus, everolimus, temsirolimus, or any other agent for current malignancy that theoretically targets Phosphoinositide 3-kinase (PI3K), AKT and / or mTOR.
* Any prior ≥ Grade 3 immune-related adverse event (irAE) while receiving immunotherapy, including anti-Cytotoxic T-Lymphocyte antigen 4 (CTLA-4) and anti-PD-1/PD-L1 treatment, or any unresolved irAE>Grade 1.

  *Note: Previous immune-related ocular toxicity of any grade is excluded.
* Subjects who are receiving an immunosuppressive treatment for any reason, including chronic use of systemic steroid or prednisone equivalent at doses ≥ 10 milligrams per day (mg/day) within 14 days prior to the first dose of study treatment. Use of inhaled or topical steroids or systemic corticosteroids < 10 mg is permitted.
* Subjects who have had prior radiotherapy within 2 weeks of therapy. Subjects must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
* Patient has received chemotherapy within 3 weeks prior to entering the study or has not recovered sufficiently (i.e., greater than grade 1. PI will judge patient recovery status) from adverse events due to agents administered more than 3 weeks earlier. Exceptions are stable chronic toxicities not expected to resolve, such as peripheral neurotoxicity, alopecia, and fatigue.
* Prior monoclonal antibody within 4 weeks before study Day 1 or not recovered (≤ Grade 1 or at baseline) from AEs due to agents administered more than 4 weeks earlier. Exception to this rule would be use of denosumab.
* Brain metastases: Symptomatic, unstable, or disease requiring use of steroid treatment.
* Subjects with any active or inactive autoimmune process (eg, rheumatoid arthritis, moderate or severe psoriasis, multiple sclerosis, inflammatory bowel disease, etc.) or who are receiving systemic therapy for an autoimmune or inflammatory disease.

  *Exceptions include subjects with vitiligo, hypothyroidism stable on hormone replacement, controlled asthma, Type I diabetes, Graves' disease, Hashimoto's disease, or with PI approval.
* Evidence of or any history of interstitial lung disease or active, noninfectious pneumonitis including symptomatic and/or pneumonitis requiring treatment.
* Hepatitis B virus (HBV) or hepatitis C virus (HCV) viremia or at risk for HBV reactivation. Hepatitis B virus deoxyribonucleic acid (DNA) and testing for HCV ribonucleic acid (RNA) must be undetectable. At risk for HBV reactivation is defined as hepatitis B surface antigen positive
* Subjects with clinical condition where subjects may not tolerate immune mediated hepatotoxicity. This includes extensive liver metastasis (See INCLUSION CRITERIA), excessive intake of alcohol (Male >4 drinks/day, Female >2 drinks>day), and the use of acetaminophen >2 gms/day. Per INCB24360 investigator's brochure.
* History or presence of an abnormal ECG which, in the investigator's opinion, is clinically meaningful. Screening corrected QT interval (QTcF) > 480ms is excluded. Subjects with left bundle branch block are excluded.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Current use or anticipated need for treatment with any medications or substances that are inhibitors or inducers of CYP3A4.
* Known allergy or reaction to any component of either study drug formulation. Any history of serotonin syndrome (SS) after receiving 1 or more serotonergic drugs.
* Pregnant or nursing. There is a potential for congenital abnormalities and for this regimen to harm nursing infants.
* Use of any UDP glucuronosyltransferase family 1 member A9 (UGT1A9) inhibitor from screening through follow-up period, including the following: diclofenac, imipramine, ketoconazole, mefenamic acid, and probenecid.
* Subjects receiving Monoamine Oxidase Inhibitors (MAOIs) or drug which has significant MAOI activity (meperidine, linezolid, methylene blue) within the 21 days before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events. | 28 days
  Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 will be used to measure incidence of treatment-emergent adverse events.

SECONDARY OUTCOMES:
Overall response response in subjects with NSCLC (dose expansion cohort) | up to 12 months
  Subjects will be assessed every 8 weeks by radiologic imaging to monitor disease status.
Disease control rate (DCR) >40% in subjects with NSCLC (dose expansion cohort) | 2 months
  Subjects will be assessed at Week 8 by radiologic imaging to monitor disease status.
Median progression free survival (mPFS) >3 months in subjects with NSCLC (dose expansion cohort) | up to 12 months
  Subjects will be assessed every 8 weeks by radiologic imaging to monitor disease status.
Median Overall Survival (mOS) > 6 months in subjects with NSCLC (dose expansion cohort) | up to 12 months
  Subjects will be assessed every 8 weeks by radiologic imaging to monitor disease status.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Huang, MD, Principal Investigator — KUMC
Locations (2):
- United States (2):
  - Clinical Research Center, Fairway, Kansas
  - The University of Kansas Cancer Center, Westwood, Kansas

IPD SHARING:
Plan to Share IPD: No